CLINICAL TRIAL: NCT06069050
Title: Sequential Adolescent Left Lateral Lobe Liver Transplantation in Adolescents With End-stage Liver Disease: a Single-center, Prospective, Single-arm Study
Brief Title: SALT in Adolescents With End-stage Liver Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LY2023-184-C
Record Dates: First submitted 2023-09-22; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: End Stage Liver DIsease
Keywords: liver transplantation; two-stage liver resection; end stage liver dIsease
MeSH Terms: conditions — End Stage Liver Disease

STUDY DESIGN:
Intervention Model Description: SALT operation plan for patients who meet the enrollment conditions and successfully match the donor liver.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgical group (Experimental): SALT operation plan for patients who meet the enrollment conditions and successfully match the donor liver: Hemihepatectomy combined with left lateral lobe liver transplantation was performed first, and residual liver resection was performed after the graft grew to a sufficient functional liver volume.
  Interventions: Procedure: sequential adolesent left lateral lobe liver transplantation (SALT)

INTERVENTIONS:
Procedure: sequential adolesent left lateral lobe liver transplantation (SALT) — Hemihepatectomy combined with left lateral lobe liver transplantation was performed first, and residual liver resection was performed after the graft grew to a sufficient functional liver volume.

SUMMARY:
End-stage liver disease is synonymous with advanced liver disease, liver failure, and decompensated cirrhosis, and their disease progression is generally irreversible. Unlike other end-stage diseases, liver transplantation is a definitive and potentially curative treatment for ESLD. However, due to clinical and social factors such as the shortage of donor livers, the number of patients who can be transplanted is far less than the number of waiting patients. About 14% of patients die each year while waiting, and about 10% of patients are too sick to be transplanted. Although changes in organ allocation policies and popularization of living donor liver transplantation have significantly reduced the waiting time and mortality of infant recipients under 2 years old. Pre-transplant mortality in children older than 6 years remains high. Therefore, expanding the donor liver pool is an urgent need to treat patients with adolescent end-stage liver disease (AESLD). In 2015, Norwegian scholars proposed a new surgical method, that is, resection and partial liver segment (2-3 segment) transplantation combined with delayed total hepatectomy can greatly alleviate the shortage of liver donors in the above patients.Based on the experience of clinical operation, our center proposes and designs the clinical research of sequential adolescent left lateral lobe liver transplantation (SALT) for the treatment of AESLD. On the basis of RAPID, the safety and efficacy of sequential juvenile left lateral lobe liver transplantation were evaluated for the above patients.

DETAILED DESCRIPTION:
Cirrhosis is an irreversible advanced stage of chronic progressive liver disease characterized by structural deformation of the liver and the formation of regenerative nodules. Those with complications are classified as decompensated cirrhosis, including variceal bleeding, ascites, spontaneous bacterial peritonitis, hepatocellular carcinoma (HCC), hepatorenal syndrome, or hepatopulmonary syndrome. These complications are the leading cause of death in patients with cirrhosis. End-stage liver disease is synonymous with advanced liver disease, liver failure, and decompensated cirrhosis, and their disease progression is generally irreversible. Unlike other end-stage diseases, liver transplantation is a definitive and potentially curative treatment for ESLD. However, due to clinical and social factors such as the shortage of donor livers, the number of patients who can be transplanted is far less than the number of waiting patients. About 14% of patients die each year while waiting, and about 10% of patients are too sick to be transplanted. Although changes in organ allocation policies and popularization of living donor liver transplantation have significantly reduced the waiting time and mortality of infant recipients under 2 years old. Pre-transplant mortality in children older than 6 years remains high. Therefore, expanding the donor liver pool is an urgent need to treat patients with adolescent end-stage liver disease (AESLD). In 2015, a new surgical method was proposed by Norwegian scholars. Therefore, expanding the donor liver pool is an urgent need to treat patients with adolescent end-stage liver disease (AESLD). In 2015, Norwegian scholars proposed a new surgical method, that is, resection and partial liver segment 2-3 transplantation with delayed total hepatectomy (RAPID). This approach allows transplantation of the left liver (segments 2+3) to an adult recipient, while the remaining enlarged right hemi-liver is transplanted to another adult recipient. Recipients who received right-hemi-liver transplantation had a similar prognosis compared with those who received whole-liver transplantation. Therefore, if the RAPID technique is confirmed to be feasible, it can greatly alleviate the shortage of liver donors. In addition to cadaver sources, living adult donors can also be considered as the source of liver donors. A smaller left lateral lobe donor liver also places less burden on the donor than a left or right hemiliver.

To sum up, our center proposed and designed a clinical study of sequential adolescent left lateral lobe liver transplantation (SALT) in the treatment of AESLD patients based on clinical surgical experience. On the basis of RAPID operation, the overall survival rate of SALT in AESLD patients was evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Age 7-18 years old;
2. Patients with end-stage liver disease cannot obtain sufficient donor liver volume through conventional living donor liver transplantation;
3. The general condition is good and can tolerate the follow-up operation plan;
4. Guardians and children (over 14 years old) sign the informed consent.

Exclusion Criteria:

1. Uncorrectable cardiopulmonary disease with excessive surgical risk
2. Anatomical abnormalities precluding liver transplantation
3. Patients with primary or secondary hepatic malignancies
4. Patients with genetic metabolic diseases and their complications that cannot be completely cured by liver transplantation
5. Persistent non-adherence to medical care
6. Combined with AIDS and other diseases that affect surgery or tumor progression
7. Other reasons that the researchers think are not suitable for participation.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-20 (Estimated); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
3-year overall survival | 3 years after the second liver resection
  To describe the 3-year overall survival after sequential adolescent left lateral lobe liver transplantation (SALT) in adolescent patients with end-stage liver disease.

SECONDARY OUTCOMES:
1-year overall survival | 1 year after the second liver resection
  To describe the 1-year overall survival after sequential adolescent left lateral lobe liver transplantation (SALT) in adolescent patients with end-stage liver disease.

IPD SHARING:
Plan to Share IPD: No